CLINICAL TRIAL: NCT04392154
Title: A Long-term Study to Assess the Safety and Efficacy of Lebrikizumab in Patients With Moderate-to-Severe Atopic Dermatitis (ADjoin)
Brief Title: Long-term Safety and Efficacy Study of Lebrikizumab (LY3650150) in Participants With Moderate-to-Severe Atopic Dermatitis (ADjoin)
Acronym: ADjoin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17789; 2020-001211-24 (EudraCT Number); J2T-DM-KGAA (Other: Eli Lilly and Company); DRM06-AD07 (Other: Dermira, Inc. (A wholly owned subsidiary of Lilly))
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lebrikizumab Q2W (Primary Treatment Period) (Experimental): 250 milligrams (mg) of Lebrikizumab, subcutaneous injection administered every 4 weeks (Q4W) up to 100 weeks.
  Interventions: Biological: Lebrikizumab
- Lebrikizumab Q4W (Primary Treatment Period) (Experimental): 250 mg Lebrikizumab, subcutaneous injection administered every 2 weeks (Q2W) up to 100 weeks.
  Interventions: Biological: Lebrikizumab
- Open-Label Extension Addendum: Lebrikizumab Q4W (Experimental): 250 mg of Lebrikizumab, subcutaneous injection administered every 4 weeks (Q4W) up to 32 weeks.
  Interventions: Biological: Lebrikizumab
- Open-Label Extension Addendum: Lebrikizumab Q8W (Experimental): 250 mg of Lebrikizumab, subcutaneous injection administered every 8 weeks (Q8W) up to 32 weeks.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150; DRM06

SUMMARY:
This is designed to assess the long-term safety and efficacy of lebrikizumab for moderate-to-severe atopic dermatitis. It will last up to 33 months.

DETAILED DESCRIPTION:
Participants who have completed participation in a Dermira- or Lilly-sponsored lebrikizumab study (parent study), DRM06-AD04 (NCT04146363), DRM06-AD05 (NCT04178967), DRM06-AD06 (NCT04250337), DRM06-AD17 (NCT04250350) or DRM06- AD18 (NCT04626297), will be offered the opportunity to enroll in this study. Participants may either be blinded or not blinded, depending on their parent study assignment.

This study will also be open to an additional approximately 100 participants in the United States (addendum) who have not completed participation in a Dermira- or Lilly-sponsored lebrikizumab study. Treatment will not be blinded.

This study will also include an Addendum to extend the study treatment period by an additional 32 weeks and to add a treatment arm testing dosing every 8 weeks. This Addendum will apply to existing study participants in selected countries. Treatment will not be blinded.

ELIGIBILITY:
Inclusion Criteria for participants coming from a parent study:

Participants must meet all the following criteria to be eligible for this study:

* Received treatment in a lebrikizumab study, NCT04146363, NCT04178967, NCT04250337, NCT04250350 and have adequately completed the study treatments and last patient visit of the parent trial.
* For women of childbearing potential: agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method during the treatment period and for at least 18 weeks after the last dose of lebrikizumab or placebo.

Exclusion Criteria for participants coming from a parent study:

Participants meeting any of the criteria below will not be included in this study:

* Participants who, during their participation in the parent trial, developed a serious adverse event (SAE) deemed related to lebrikizumab, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with lebrikizumab may present an unreasonable risk for the participant. *
* Participants who, during their participation in the parent trial, developed an AE that was deemed related to lebrikizumab and led to study treatment discontinuation, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with lebrikizumab may present an unreasonable risk for the participant. *
* Conditions in the previous parent study consistent with protocol-defined criteria for permanent study drug discontinuation, if deemed related to lebrikizumab or led to investigator - or sponsor-initiated withdrawal of participant from the study (e.g., non-compliance, inability to complete study assessments, etc.). *
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Open-Label Addendum Inclusion Criteria:

Participants must meet all the following criteria to be eligible for this study addendum:

* Male or female adults and adolescents (≥12 to <18 years of age and weighing ≥40 kilogram (kg).
* Chronic AD (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before screening.
* Eczema Area and Severity Index (EASI) score ≥16 at baseline.
* Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at baseline.
* ≥10% body surface area (BSA) of AD involvement at baseline.
* History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.

Open-Label Addendum Exclusion Criteria:

Participants meeting any of the criteria below will be excluded from this study addendum:

* Have received a dose of lebrikizumab in any prior lebrikizumab clinical study.
* History of anaphylaxis
* Treatment with topical prescription moisturizers, corticosteroids, calcineurin inhibitors, or phosphodiesterase-4 inhibitors such as crisaborole within 1 week prior to baseline.
* Treatment with any of the following agents within 4 weeks prior to the baseline.

  * Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, Interferon gamma (IFN-γ), Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  * Phototherapy and photochemotherapy (PUVA) for AD.
* Treatment with the following prior to baseline:

  * Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  * Phototherapy and photochemotherapy (PUVA) for AD.
* Treatment with the following prior to baseline:

  * An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer.
  * B Cell-depleting biologics, including rituximab, within 6 months.
  * Other Biologics within 5 half-lives (if known) or 8 weeks, whichever is longer.
* Regular use (more than 2 uses per week) of a tanning booth/parlor within 4 weeks of baseline.
* Treatment with a live (attenuated) vaccine within 12 weeks of the baseline or planned during the study.
* Uncontrolled chronic disease that might require multiple intermittent uses of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma, (as defined by the investigator).
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
* Evidence of active acute or chronic hepatitis
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* History of malignancy, including mycosis fungoides, within 5 years before screening, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.

Open-Label Extension Addendum Inclusion Criteria:

Have completed Week 100 of Study KGAA and have not yet completed the safety follow-up visit for the main study.

Open-Label Extension Addendum Exclusion Criteria:

Have initiated treatment with a medication prohibited by Study KGAA before addendum baseline. This includes use of biologics for AD (for example, dupilumab and tralokinumab) during the safety follow-up period of Study KGAA.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (317):
- United States (159):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Clinical Research Center of Alabama- Birmingham, Birmingham, Alabama
  - Investigate MD, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Wallace Medical Group, Inc., Beverly Hills, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - MD Studies, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Axon Clinical Research, Inglewood, California
  - Sunwise Clinical Research, Lafayette, California
  - Avance Clinical Trials Inc, Laguna Niguel, California
  - California Allergy and Asthma Medical Group + Research Center, Los Angeles, California
  - Keck School of Medicine University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - LA Universal Research Center, INC, Los Angeles, California
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Dermatology Clinical Trials, Newport Beach, California
  - Cura Clinical Research, Palmdale, California
  - MD Strategies Research Centers MDSRC, Poway, California
  - Integrative Skin Science and Research, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - University Clinical Trials, San Diego, California
  - University of California, San Diego/Rady Children's Hospital, San Diego - Pediatric & Adolescent Dermatology, San Diego, California
  - Synergy Dermatology, San Francisco, California
  - Care Access Research, San Jose, California
  - San Luis Dermatology & Laser Clinic, San Luis Obispo, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Central Connecticut Dermatology, Cromwell, Connecticut
  - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Pediatric Skin Research, LLC, Coral Gables, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - The University of Florida Health System, Gainesville, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - GSI Clinical Research, LLC, Margate, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Community Research Foundation Inc, Miami, Florida
  - Sanchez Clinical Research Inc, Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Florida Research Center, Inc, Miami, Florida
  - C & R Research Services USA, Miami Beach, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc, Albany, Georgia
  - IACT Health - VHC, Columbus, Georgia
  - Marietta Dermatology Clinical Research, Marietta, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates LLC, Normal, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Kansas Medical Clinic, an Elligo Health Research, Inc., Shawnee Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Tulane Univ School of Med, New Orleans, Louisiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - ActivMed Practices and Research, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Fivenson Dermatology, Ann Arbor, Michigan
  - Oakland Dermatology, Auburn Hills, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Michigan Center for Research Company, Clarkston, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - Associated Skin Care Specialists, Fridley, Minnesota
  - Associated Skin Care Specialists, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Central Dermatology PC, St Louis, Missouri
  - Advanced Dermatology of the Midlands, Omaha, Nebraska
  - JDR Dermatology Research, Las Vegas, Nevada
  - ALLCUTIS Research, Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Skin Laser and Surgery Specialists, a Division of Schweiger Dermatology, Hackensack, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - JUVA Skin & Laser Center, New York, New York
  - Icahn Sch of Med at Mt. Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Advanced Asthma and Allergy, Watertown, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Crisor, LLC, Medford office, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - DermDox Dermatology Centers, Sugarloaf, Pennsylvania
  - Peak Research LLC, Upper Saint Clair, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - Palmetto Clinical Trial Services, LLC, Anderson, South Carolina
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Rivergate Dermatology Clinical Research Center PL, Goodlettsville, Tennessee
  - Arlington Research Center, Inc, Arlington, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Austin Institute for Clinical Research, Dripping Springs, Texas
  - Innovate Research, LLC, Fort Worth, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Encore Imaging & Medical Research, Houston, Texas
  - Cutis Wellness Dermatology, Laredo, Texas
  - Laredo Dermatology Associates P.A., Laredo, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Acclaim Dermatology PLLC, Sugar Land, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Velocity Clinical Research - Woseth Dermatology, Salt Lake City, Utah
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Australia (19):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - The Skin Hospital, Darlinghurst, New South Wales
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - The St. George Hospital, Kogarah, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - University of the Sunshine Coast Clinical Trial Centre, Sippy Downs, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Clinical Trials SA Pty Ltd, Hectorville, South Australia
  - Emeritus Research, Camberwell, Victoria
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Burswood Dermatology, Victoria Park, Western Australia
  - Captain Stirling Medical Centre, Nedlands
- Bulgaria (6):
  - DCC Sveti Georgi, Haskovo
  - Diagnostic and Consultation Center 14, Sofia
  - Alexandrovska University Hospital, Sofia
  - Euro Derma clinic, Sofia
  - Military Medical Academy, Sofia
  - Medical centre Alitera-Med EOOD, Sofia
- Canada (19):
  - Dermatology Research Institute, Calgary, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - CCA Medical Research, Ajax, Ontario
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Skin Health, Cobourg, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North York Research Inc., North York, Ontario
  - The Centre for Clinical Trials, Inc, Oakville, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - Skin Health, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - AvantDerm, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - International Dermatology Research, Montreal, Quebec
- Estonia (3):
  - Vahlberg & Pild OU, Talinn
  - Kliiniliste uuringute Keskus OU, Tartu
  - Tartu University Hospital, Tartu
- France (9):
  - CHU de Bordeaux Hop St ANDRE, Bordeaux, Gironde
  - CHRU de Brest - Hôpital Morvan, Brest
  - CHU Dijonon, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - Cabinet Médical, Martigues
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - CHU de Nice Hopital de L'Archet, Nice
  - Hopital Saint Louis, Paris
  - Hopital Larrey, Toulouse
- Germany (22):
  - Studienzentrum Dr.Beate Schwarz, Langenau, Baden-Wurttemberg
  - Hautarztpraxis am Löwenmarkt, Stuttgart, Baden-Wurttemberg
  - Dermazentrum Augsburg, Augsburg, Bavaria
  - Rosenpark Research GmbH, Darmstadt, Hesse
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Elbe Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Klinische Forschung Osnabrück, Osnabrück, Lower Saxony
  - Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Company for Medical Study & Service Selters GmbH, Selters, Rhineland-Palatinate
  - Hautarztpraxis Dr. Gerlach, Dresden, Saxony
  - Technische Universitaet Dresden - Universitaetsklinikum Carl Gustav Carus - Klinik und Poliklinik fuer, Dresden, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Velocity Clinical Research Leipzig GmbH, Leipzig, Saxony
  - SRH Wald-Klinikum Gera, Gera, Thuringia
  - Praxis Dr. med. Virgil-Oreste Mihaescu Facharzt fr Dermatologie und STD, Augsburg
  - Charité Campus Virchow-Klinikum, Berlin
  - ISA GmbH, Berlin
  - Praxis für Ganzheitliche Dermatologie im Ärztehaus, Berlin
  - Dermatologikum Hamburg, Hamburg
  - TFS Trial Support Form GmbH, Hamburg
- Latvia (5):
  - Clinic of Dermatology and STD, Riga
  - Health and Aesthetics LTD, Riga
  - Latvian Dermatology Institute, Riga
  - Health Center 4, Affiliate Diagnostic Center, Riga
  - Smite Aija - Doctor Practice in Dermatology Venereology, Talsi
- Lithuania (7):
  - JSC "CD8 Alergology Clinic", Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Children's Hospital, Affiliate of Vilnius University Hospital Santaros klinikos, Vilnius
  - Jsc Renmeda, Vilnius
  - JSC "Center for Diagnosis and Treatment of Allergic Diseases", Vilnius
  - JSC Inlita (Santaros CTC), Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (6):
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Federal District
  - Grupo Clinico CATEI Sociedad Civil, Guadalajara, Jalisco
  - Clinica De Enfermedades Cronicas y Procedimientos Especiales, Morelia, Michoacán
  - Cemdeicy S.C.P., Mérida, Yucatán
  - Derma Norte del Bajio, Aguascalientes
  - Arke Estudios Clinicos S.A. de C.V., Veracruz
- Poland (27):
  - Grazyna Pulka Specjalistyczny Osrodek "ALL-MED", Krakow, Lesser Poland Voivodeship
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - dermMedica Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Centralny Szpital Kliniczny MSWiA, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Zespol Naukowo - Leczniczy "Iwolang" Sp. z o.o., Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Labderm s.c., Ossy, Silesian Voivodeship
  - Laser Clinic Dermatologia Laserowa Medycyna Estetyczna, Szczecin, West Pomeranian Voivodeship
  - Clinica Vitae Sp. z o.o., Gdansk, Woj. Pomorskie
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny Anna Ploszczuk, Bialystok
  - Wojewodzki Szpital Zespolony, Elblag
  - Oddzial Dermatologii COPERNICUS, Gdansk
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdynia
  - Holsamed, Katowice
  - Gabinet Dermatlogiczny. Beata Krecisz, Kielce
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - Kliniczny Szpital Wojewodzki nr. 1 Klinika Dermatologii, Rzeszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp Z O.O., Tarnów
  - Clinical Research Group Sp. z o.o., Warsaw
  - High-Med Prywatny Gabinet Lekarski, Warsaw
  - MTZ Clinical Research Sp.z.o.o., Warsaw
  - Klinika Ambroziak Sp. Z.O.O., Warsaw
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
  - Dermoklinika Centrum Medyczne s.c. M. Kierstan J. Narbutt A. Lesiak, Lodz, Łódź Voivodeship
- Singapore (4):
  - National University Hospital, Singapore, Central Singapore
  - Singapore General Hospital, Singapore
  - Kk Women'S and Childrens Hospital, Singapore
  - National Skin Centre NSC, Singapore
- South Korea (11):
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Pusan National University Hospital, Busan, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Ansan Hospital, Gyeonggi-do
  - Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (8):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Hospital Germans Trias i Pujol, Badalona, Catalunya [Cataluña]
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Basurto, Bilbao (Bizkaia)
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Niaosong, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- Ukraine (5):
  - Community Institution Zaporizhzhya Regional Dermatovenereology Clinical Hospital of Zaporizhzhya Regional Council, Poshtova Square 2, Zaporizhzhya
  - Municipal Healthcare Institution Kharkiv City Dermatoverenologic Dispensary N2, Kharkiv
  - SE "Institute of Dermatology and Venerology of NAMS of Ukraine", Kharkiv
  - Rivne Regional Dermatology and Venereology Dispensary, Rivne
  - Treatment-diagnostic center PE "Asclepius", Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Silverberg JI, Wollenberg A, Stein Gold L, Yosipovitch G, Lio P, Vestergaard C, Stander S, Carrascosa JM, Gallo G, Casillas M, Ding Y, Yang FE, Pierce E, Agell H, Del Rosso J. Lebrikizumab provides stable skin response with no or minimal fluctuations for up to 2 years in patients with atopic dermatitis. Clin Exp Dermatol. 2025 Nov 8:llaf490. doi: 10.1093/ced/llaf490. Online ahead of print. PMID 41206702
- [Derived] Guttman-Yassky E, Weidinger S, Simpson EL, Gooderham M, Irvine AD, Spelman L, Silverberg JI, ElMaraghy H, DeLuca-Carter L, Piruzeli MLB, Hu C, Yang FE, Pierce E, Bardolet L, Thaci D. Two-Year Efficacy and Safety of Lebrikizumab in Patients with Moderate-to-Severe Atopic Dermatitis: A Long-Term Extension (ADjoin). Dermatol Ther (Heidelb). 2025 Aug;15(8):2217-2232. doi: 10.1007/s13555-025-01452-9. Epub 2025 Jun 23. PMID 40549127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consists of 2 parts:
  * 100-week primary treatment period where participants were assigned to either Lebrikizumab Q4W or Q2W treatment arms.
  * 32-week open label extension addendum (Lebrikizumab Q4W and Lebrikizumab Q8W)
Groups:
- Primary Treatment Period: Lebrikizumab Q4W: 250 milligrams (mg) of Lebrikizumab, subcutaneous injection administered every 4 weeks (Q4W) up to 100 weeks.
- Primary Treatment Period: Lebrikizumab Q2W: 250 mg Lebrikizumab, subcutaneous injection administered every 2 weeks (Q2W) up to 100 weeks.
Period: Primary Treatment Period (100 Weeks)
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W | Open-Label Extension Addendum: Lebrikizumab Q4W | Open-Label Extension Addendum: Lebrikizumab Q8W
Started | 141 | 1012 | 0 | 0
Received at Least 1 Dose of Study Drug | 141 | 1012 | 0 | 0
Completed | 103 | 675 | 0 | 0
Not Completed | 38 | 337 | 0 | 0
Not completed — Adverse Event | 3 | 46 | 0 | 0
Not completed — Due to epidemic/pandemic | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 47 | 0 | 0
Not completed — Lost to Follow-up | 11 | 61 | 0 | 0
Not completed — Geopolitical conflict | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 5 | 0 | 0
Not completed — Pregnancy | 1 | 8 | 0 | 0
Not completed — Protocol deviation | 1 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 138 | 0 | 0
Not completed — Sponsor Decision | 1 | 14 | 0 | 0
Not completed — Site Closure | 0 | 4 | 0 | 0
Period: Open-Label Extension Addendum (32 Weeks)
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W | Open-Label Extension Addendum: Lebrikizumab Q4W | Open-Label Extension Addendum: Lebrikizumab Q8W
Started | 0 | 0 | 52 (Participants who completed the 100-week primary treatment period, regardless of their previous treatment regimen (Lebrikizumab Q2W or Q4W), had the option to enter the open-label extension addendum to receive Lebrikizumab 250 mg Q4W or Q8W.) | 51 (Participants who completed the 100-week primary treatment period, regardless of their previous treatment regimen (Lebrikizumab Q2W or Q4W), had the option to enter the open-label extension addendum to receive Lebrikizumab 250 mg Q4W or Q8W.)
Received at Least One Doe of Study Drug | 0 | 0 | 52 | 51
Completed | 0 | 0 | 51 | 49
Not Completed | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Primary Treatment Period: Lebrikizumab Q4W: 250 mg of Lebrikizumab, subcutaneous injection administered every 4 weeks (Q4W) up to 100 weeks.
- Total: Total of all reporting groups
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W | Total
Number analyzed (Participants) | 141 | 1012 | 1153
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (16.96) | 32.5 (17.23) | 32.8 (17.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 513 | 595
  Male | 59 | 499 | 558
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 16 | 17
  Asian | 21 | 199 | 220
  Native Hawaiian or Other Pacific Islander | 1 | 9 | 10
  Black or African American | 9 | 138 | 147
  White | 106 | 610 | 716
  More than one race | 3 | 25 | 28
  Unknown or Not Reported | 0 | 15 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 1 | 7 | 8
  United States | 72 | 591 | 663
  Ukraine | 5 | 4 | 9
  Spain | 0 | 7 | 7
  Canada | 14 | 80 | 94
  Latvia | 3 | 5 | 8
  South Korea | 2 | 25 | 27
  Taiwan | 4 | 51 | 55
  Poland | 23 | 135 | 158
  Mexico | 2 | 2 | 4
  Australia | 3 | 23 | 26
  Bulgaria | 0 | 10 | 10
  France | 1 | 3 | 4
  Lithuania | 1 | 12 | 13
  Germany | 10 | 52 | 62
  Estonia | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Treatment Period: Percentage of Participants Discontinued From Study Treatment Due to Adverse Events
Description: Percentage of participants discontinued from study treatment due to adverse events is reported.
Time Frame: Baseline to Week 100
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 1012
percentage of participants | 2.1 | 4.5

2. Secondary Outcome: Primary Treatment Period: Percentage of Participants With a Response of Investigator Global Assessment (IGA) Score 0 or 1 at Week 100
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their Atopic Dermatitis. The IGA is comprised of a 5-point numeric scale ranging from 0 (clear skin) to 4 (severe disease) and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point.
Time Frame: Week 100
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 1012
Percentage of participants | 80.1 | 60.6

3. Secondary Outcome: Primary Treatment Period: Percentage of Participants Achieving Response of Eczema Area and Severity Index-75 (EASI-75) at Week 100
Description: EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs, by scoring the extent of disease (percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed. The final EASI score will be obtained by weight-averaging these 4 scores and will range from 0 to 72. A higher score represents greater disease severity.
Time Frame: Week 100
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W
Number analyzed (Participants) | 141 | 1012
Percentage of participants | 90.4 | 79.4

ADVERSE EVENTS:
Time Frame: Primary Treatment Period: Up to 110 Weeks; Open-Label Extension Addendum: up to 42 weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Primary Treatment Period: Lebrikizumab Q4W | Primary Treatment Period: Lebrikizumab Q2W | Open-Label Extension Addendum: Lebrikizumab Q4W | Open-Label Extension Addendum: Lebrikizumab Q8W
All-Cause Mortality (participants affected / at risk) | 0/141 | 2/1012 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 5/141 | 45/1012 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 89/141 | 638/1012 | 17/52 | 13/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Treatment Period: Lebrikizumab Q4W (N=141) | Primary Treatment Period: Lebrikizumab Q2W (N=1012) | Open-Label Extension Addendum: Lebrikizumab Q4W (N=52) | Open-Label Extension Addendum: Lebrikizumab Q8W (N=51)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden visual loss (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Treatment Period: Lebrikizumab Q4W (N=141) | Primary Treatment Period: Lebrikizumab Q2W (N=1012) | Open-Label Extension Addendum: Lebrikizumab Q4W (N=52) | Open-Label Extension Addendum: Lebrikizumab Q8W (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 10 (12) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 9 (10) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Polycystic ovarian syndrome (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Blepharitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 29 (39) | 0 (0) | 0 (0)
Corneal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Keratoconus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital dermatitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 13 (15) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal vascular disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Malpositioned teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 9 (10) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 12 (32) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 8 (16) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metabolic dysfunction-associated liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic dysfunction-associated steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to venom (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dust allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 9 (10) | 0 (0) | 0 (0)
Abscess of eyelid (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (3) | 1 (4) | 0 (0) | 0 (0)
Blastocystis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 11 (11) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (4) | 39 (45) | 1 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 26 (29) | 159 (172) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythrasma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (3) | 11 (12) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 13 (16) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 2 (3) | 10 (15) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 11 (15) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 2 (3) | 8 (10) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 12 (12) | 0 (0) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malassezia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (14) | 115 (165) | 2 (2) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (3) | 30 (46) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 15 (15) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Toxocariasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (11) | 49 (63) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 30 (35) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 5 (10) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 17 (18) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (8) | 0 (0) | 0 (0)
Bilirubin urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood immunoglobulin e increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Double stranded dna antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin urine present (Investigations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte morphology abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Red blood cell morphology abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Treponema test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Histamine intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Periarthritis calcarea (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 15 (19) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 14 (17) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 25 (33) | 1 (1) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 11 (11) | 0 (0) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar i disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 10 (10) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (26) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 12 (13) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 17 (19) | 1 (1) | 0 (0)
Acne varioliformis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (8) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 (12) | 70 (102) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lichen striatus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (9) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (11) | 0 (0) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 15 (15) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accessory navicular syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT04392154/Prot_000.pdf
  • Study Protocol: Study Protocol Addendum (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04392154/Prot_002.pdf
  • Statistical Analysis Plan (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT04392154/SAP_001.pdf